CLINICAL TRIAL: NCT01788358
Title: Multicenter, Open-Label, Long-Term Safety and Efficacy Study of the Fixed Dose Combination of Nifedipine Gastrointestinal Therapeutic System and Candesartan Cilexetil in Adult Subjects With Moderate to Severe Essential Hypertension
Brief Title: Open-Label Long-Term Safety and Efficacy Study of Fixed Dose Combination of Nifedipine Gastrointestinal Therapeutic System and Candesartan Cilexetil in Subjects With Moderate to Severe Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14801; 2012-004515-32 (EudraCT Number)
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-09

CONDITIONS: Hypertension
Keywords: Drug combination; Nifedipine GITS; Candesartan Cilexetil; Hypertension; Combination therapy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106) (Experimental): Subjects received nifedipine gastrointestinal therapeutic system (GITS) / candesartan cilexetil fixed dose combination (FDC) (BAY98-7106) tablet orally, once daily in the morning of Visit 1 (Week 0) for 28 or 52 weeks. The starting dose (30/8 milligram [mg] or 30/16 mg) was determined based on local practice and clinical judgment by the investigator. Based on the experience of symptomatic and asymptomatic hypotension, peripheral edema or significant tolerability, the doses were up-titrated to the highest target dose (60/32 mg).
  Interventions: Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106)

INTERVENTIONS:
Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) — Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106), tablet, 30/8 mg, orally once daily
Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) — Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106), tablet, 30/16 mg, orally once daily
Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) — Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106), tablet, 60/16 mg, orally once daily
Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) — Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106), tablet, 60/32 mg, orally once daily

SUMMARY:
This study examines the long term safety and efficacy of the Fixed Dose combination BAY98-7106 (nifedipine plus candesartan primarily at the highest dose in development) in patients with moderate to severe hypertension.

Patients meeting the entry criteria, will receive the Fixed Dose combination for 28 weeks, including 8 weeks with stepwise dose increase up to the high target dose. The first 200 subjects completing 28 weeks will continue treatment for additional 24 weeks (52 weeks in total).

Subjects who do not tolerate an increased dose will be treated at their highest tolerable dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have moderate to severe essential hypertension (Grade 2 or Grade 3, WHO classifications). At Visit 1, subjects not treated with antihypertensive medications are to have MSSBP of >/= 160 mmHg and < 200 mmHg, as measured by a calibrated electronic BP measuring device. For other subjects who are treated with antihypertensive medication before, they should have MSSBP >/= 160 mmHg and <200 mmHg after wash out.
* Women of childbearing potential and men must agree to use adequate contraception other than hormonal contraceptives when sexually active

Exclusion Criteria:

* Mean seated systolic blood pressure >/= 200 mmHg and/or mean seated diastolic blood pressure >/= 120 mm/Hg
* Mean seated diastolic blood pressure < 60 mm/Hg
* Differences greater than 20 mmHg for systolic blood pressure and 10 mmHg for diastolic blood pressure are present on 3 consecutive blood pressure readings at visit 0
* Any history of hypertensive emergency
* Evidence of secondary hypertension such as coarctation of the aorta, pheochromocytoma, hyperaldosteronism, etc.
* Cerebrovascular ischemic event (stroke, transient ischemic attack [TIA])within the previous 12 months
* History of intracerebral hemorrhage or subarachnoid hemorrhage
* History of hypertensive retinopathy - known Keith-Wagener Grade III or IV
* Any history of heart failure, New York Heart Association (NYHA) classification III or IV
* Severe coronary heart disease as manifest by a history of myocardial infarction or unstable angina in the last 6 months prior to visit 0
* Type 1 diabetes mellitus (DM) or poorly controlled Type 2 DM as evidenced by HbA1C of greater than 9% on visit 0.
* Hyperkalemia: potassium above the upper limit of normal in the laboratory range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2013-02-14 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2014-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (78):
- United States (36):
  - Foley, Alabama
  - Carmichael, California
  - Los Angeles, California
  - Spring Valley, California
  - Milford, Connecticut
  - Coral Gables, Florida
  - Hallandale, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Valparaiso, Indiana
  - Newton, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Auburn, Maine
  - Elkridge, Maryland
  - Brockton, Massachusetts
  - St Louis, Missouri
  - Shelby, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Greenville, South Carolina
  - Mt. Pleasant, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - New Tazewell, Tennessee
  - Beaumont, Texas
  - Bryan, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Kenosha, Wisconsin
- Belgium (5):
  - Moorsel, Oost-Vlaanderen
  - Wetteren, Oost-Vlaanderen
  - Steenokkerzeel, Vlaams Brabant
  - Deurne
  - Ham
- Canada (14):
  - Burnaby, British Columbia
  - Langley, British Columbia
  - Vancouver, British Columbia
  - Brampton, Ontario
  - Burlington, Ontario
  - Etobicoke, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Sarnia, Ontario
  - Stayner, Ontario
  - Toronto, Ontario
  - Woodstock, Ontario
  - Pointe-Claire, Quebec
  - Ste-Foy, Quebec
- Germany (7):
  - Frankfurt am Main, Hesse
  - Bochum, North Rhine-Westphalia
  - Görlitz, Saxony
  - Leipzig, Saxony
  - Magdeburg, Saxony-Anhalt
  - Berlin
  - Dresden
- Poland (4):
  - Gdynia
  - Katowice
  - Warsaw
  - Wroclaw
- United Kingdom (12):
  - Reading, Berkshire
  - Chesterfield, Derbyshire
  - Blackpool, Lancashire
  - Bath, Somerset
  - Bury Saint Edmonds, Suffolk
  - Coventry, Warwickshire
  - Birmingham, West Midlands
  - Cardiff
  - Chorley
  - Glasgow
  - Liverpool
  - Manchester

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 70 study centers between 14 February 2013 (first subject first visit) and 1 May 2014 (last subject last visit).
Pre-assignment Details: Of 753 subjects screened, 245 subjects were not enrolled, due to screen failure for 215 subjects, consent withdrawal by 23 subjects, protocol violation by 5 subjects, 1 subject was lost to follow-up and recruitment stopped for 1 subject. Remaining 508 subjects were enrolled and received at least 1 treatment with study drug.
Period: Overall Study
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Started | 508
Treated | 508
Completed Week 28 | 417
Entered Extension to Week 52 | 200 (Only the first 200 subjects who completed Week 28 visit, continued treatment up to 52 weeks.)
Completed Week 52 | 193
Completed | 410 (217 subjects completed the study at Week 28 while the remaining 193 subjects completed at Week 52)
Not Completed | 98
Not completed — Other | 11
Not completed — Logistical difficulties | 1
Not completed — Lost to Follow-up | 5
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 26
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 51

BASELINE CHARACTERISTICS:
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Number analyzed (Participants) | 508
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186
  Male | 322
Systolic blood pressure [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 170.7 (8.9)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 95.6 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With All Treatment-emergent Adverse Events (TEAEs) and Drug-related TEAEs up to Week 28
Description: An adverse event (AE) is any untoward medical occurrence (that is, any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study. AEs were considered to be treatment-emergent if they had started or worsened after first application of study medication.
Time Frame: From the time of first study drug administration up to Week 28
Population: Safety Analysis Set (SAF): All the subjects enrolled into the open-label treatment period and took at least one unit of the study medication.
Measure: Number; unit: Subjects
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Number analyzed (Participants) | 508
Subjects
  All TEAEs | 390
  Drug-related TEAEs | 230

2. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs) of Special Interest up to Week 28
Description: An AE is any untoward medical occurrence (that is, any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study. AEs were considered to be treatment-emergent if they had started or worsened after first application of study medication. TEAEs of special interest included the incidence of symptomatic hypotension and the incidence and severity of vasodilatory adverse events (such as oedema, headache, and flushing). Only subjects who had TEAEs of special interest as mild, moderate or severe were reported.
Time Frame: From the time of first study drug administration up to Week 28
Population: SAF
Measure: Number; unit: Subjects
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Number analyzed (Participants) | 508
Subjects
  Oedema (mild) | 124
  Oedema (moderate) | 54
  Oedema (severe) | 7
  Headache (mild) | 31
  Headache (moderate) | 15
  Flushing (mild) | 3
  Symptomatic hypotension (mild) | 4

3. Primary Outcome: Number of Subjects With All Treatment-emergent Adverse Events (TEAEs) and Drug-related TEAEs up to Week 52/End of Study (EOS)
Description: An AE is any untoward medical occurrence (that is, any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study. AEs were considered to be treatment-emergent if they had started or worsened after first application of study medication.
Time Frame: From the time of first study drug administration up to Week 52/EOS
Population: SAF
Measure: Number; unit: Subjects
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Number analyzed (Participants) | 508
Subjects
  All TEAEs | 404
  Drug-related TEAEs | 238

4. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs) of Special Interest up to Week 52/End of Study (EOS)
Description: as for outcome 2
Time Frame: From the time of study treatment up to Week 52/EOS
Population: SAF
Measure: Number; unit: Subjects
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Number analyzed (Participants) | 508
Subjects
  Oedema (mild) | 131
  Oedema (moderate) | 56
  Oedema(severe) | 7
  Headache (mild) | 31
  Headache (moderate) | 17
  Flushing (mild) | 3
  Symptomatic hypotension (mild) | 4

5. Secondary Outcome: Number of Subjects With Clinically Relevant Changes in Laboratory Parameters
Description: Laboratory evaluations of blood and urine samples were performed, including hematology (hematocrit, hemoglobin, red blood cells count, white blood cells count, neutrophils, lymphocytes, monocytes, eosinophils, basophils, platelets), blood chemistry (sodium, potassium, chloride, bicarbonate, uric acid, total protein, albumin, calcium, blood urea nitrogen, creatinine, aspartate transaminase, alanine transaminase, lactate dehydrogenase, gamma glutamyl transferase, alkaline phosphatase, creatine kinase, total bilirubin, direct bilirubin, total cholesterol, low density lipoprotein cholesterol, high density lipoprotein cholesterol, triglycerides, fasting glucose), urinalysis (pH, blood, specific gravity, glucose, protein, cells/sediment). A laboratory test abnormality considered clinically relevant, for example, causing withdrawal by subject, requiring treatment or causing apparent clinical manifestations, or judged relevant by the investigator, were reported as AEs.
Time Frame: Baseline (Week 0) up to Week 52/EOS
Population: SAF
Measure: Number; unit: Subjects
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Number analyzed (Participants) | 508
Subjects | 0

6. Secondary Outcome: Change From Baseline In Mean Seated Systolic Blood Pressure (MSSBP) At Weeks 28 And 52
Time Frame: Baseline (Week 0), Weeks 28 and 52
Population: Modified intention-to-treat analysis set (mITT): All the subjects enrolled into the open-label treatment period and took at least one unit of the study medication.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Number analyzed (Participants) | 508
millimeter of mercury (mmHg)
  Baseline | 170.7 (8.9) [lower limit 8.9]
  Change at Week 28 | -30.4 (17.7) [lower limit 17.7]
  Change at Week 52 | -30.1 (18.4) [lower limit 18.4]

7. Secondary Outcome: Change From Baseline in Mean Seated Diastolic Blood Pressure (MSDBP) at Weeks 28 and 52
Time Frame: Baseline (Week 0), Weeks 28 and 52
Population: mITT
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Number analyzed (Participants) | 508
millimeter of mercury (mmHg)
  Baseline | 95.6 (10.4) [lower limit 10.4]
  Change at Week 28 | -12.7 (10.6) [lower limit 10.6]
  Change at Week 52 | -12.8 (10.7) [lower limit 10.7]

8. Secondary Outcome: Blood Pressure Control Rate at Weeks 28 and 52
Description: Control rate was defined as the percentage of subjects that reached a predetermined blood pressure (BP) target of BP less than (<) 140/90 mmHg.
Time Frame: Weeks 28 and 52
Population: mITT
Measure: Number; unit: percentage of subjects
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Number analyzed (Participants) | 508
percentage of subjects
  Week 28 | 51.4
  Week 52 | 51.6

9. Secondary Outcome: Blood Pressure Response Rate at Weeks 28 and 52
Description: Response rate was defined as the percentage of subjects who achieved a systolic blood pressure response (MSSBP of <140 mmHg or a reduction of MSSBP of more than (>) 20 mmHg from baseline value), or a diastolic blood pressure response (MSDBP of <90 mmHg or a reduction of MSDBP of >10 mmHg from baseline value).
Time Frame: Weeks 28 and 52
Population: mITT
Measure: Number; unit: percentage of subjects
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Number analyzed (Participants) | 508
percentage of subjects
  Week 28 | 86.6
  Week 52 | 86.2

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) were collected from the time of first study drug administration up to 7 days after Week 52/EOS
Description: One death reported under SAE happened approximately 6 months after the subject had completed the study due to malignant melanoma of head and neck with metastasis to lung and liver, not related to the treatment.
Arm/Group | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106)
Serious Adverse Events (participants affected / at risk) | 15/508
Other Adverse Events (participants affected / at risk) | 279/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106) (N=508)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nifedipine GITS/Candesartan Cilexetil FDC (BAY98-7106) (N=508)
Fatigue (General disorders) | 18 (20)
Oedema (General disorders) | 55 (80)
Oedema peripheral (General disorders) | 150 (239)
Nasopharyngitis (Infections and infestations) | 27 (30)
Upper respiratory tract infection (Infections and infestations) | 25 (29)
Dizziness (Nervous system disorders) | 47 (55)
Headache (Nervous system disorders) | 47 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less